CLINICAL TRIAL: NCT05888389
Title: Safety of Nerve Block Anesthesia Combined With Sedative Anesthesia Versus General Anesthesia in Burr Hole Craniostomy With Drainage for Chronic Subdural Hematoma
Brief Title: Nerve Block Anesthesia Combined With Sedative Anesthesia Versus General Anesthesia in Surgery for CSDH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Weiming Liu, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-B-2022078
Record Dates: First submitted 2023-05-07; First posted 2023-06-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Chronic Subdural Hematoma; Anesthesia
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (GA) (Active Comparator): The GA group will receive general anesthesia.
  Interventions: Procedure: General Anesthesia
- Cranial nerve block anesthesia combined with sedative anesthesia (CNB-D) (Experimental): The CNB-D group will receive cranial nerve block anesthesia combined with sedative anesthesia
  Interventions: Procedure: Cranial Nerve Block Anesthesia Combined With Sedative Anesthesia

INTERVENTIONS:
Procedure: Cranial Nerve Block Anesthesia Combined With Sedative Anesthesia — Patients in the nerve block anesthesia combined with sedative anesthesia group will first receive cranial nerve blocks under standard monitoring. At the same time, intravenous dexmedetomidine infusion is started for sedation at a rate of 2-4ug/kg for 10 minutes, followed by a continuous infusion of 0.5-1ug/kg/h until the Richmond Agitation-Sedation Scale (RASS) of -3.
  Arms: Cranial nerve block anesthesia combined with sedative anesthesia (CNB-D)
Procedure: General Anesthesia — Patients will be induced with propofol or etomidate, sufentanil , rocuronium or cisatracurium .
  Arms: General anesthesia (GA)

SUMMARY:
A prospective, multicenter, randomized controlled trial is designed to evaluate the safety of nerve block anesthesia combined with sedative anesthesia versus general anesthesia during burr hole craniostomy with drainage for chronic subdural hematoma.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, randomised, controlled, single-blinded, non-inferiority trial. Patients with chronic subdural hematoma undergoing burr-hole drainage will be randomly allocated to receive either the cranial nerve block with dexmedetomidine sedation or general anaesthesia. Patients in the cranial nerve block with dexmedetomidine sedation group will receive cranial nerve block with 0.5% ropivacaine and 1% lidocaine mixture according to incision, combined with dexmedetomidine infusion at a rate of 2-4ug/kg for 10 minutes, followed by a continuous infusion of 0.5 to 1ug/kg/h until the end of the operation. Patients in the general anaesthesia group will be induced with propofol or etomidate, sufentanil, rocuronium or cis-atracurium and be maintained with total intravenous anaesthesia. The primary outcome is the incidence of intraoperative limb movement. Secondary outcomes include postoperative delirium within five days after surgery, anaesthesia conversion, postoperative neurological function, intraoperative awareness, and recurrence rate of hematoma within 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic subdural hematoma with preoperative neurological dysfunction for burr hole drainage;
* Age beween 18 to 80
* Chronic subdural hematoma verified on cranial computed tomography or magnetic resonance imaging with hematoma thickness >1.0cm or midline shift >1.0 cm.
* Written informed consent obtained

Exclusion Criteria:

* Preoperative unconsciousness (Glasgow Coma Scale<13, or Markwalder Grade 2-4) or cognitive dysfunction (Mini-Cog≤3, or MMSE≤20)
* Preoperative sensory or motor aphasia
* Recurrence of hematoma with previous surgery for chronic subdural hematoma.
* Previous intracranial surgery or with intracranial lesion
* with severe comorbidity or other organ dysfunction
* Allergic to anesthetics
* Severe coagulopathy or high risk of life-threatening bleeding
* Participating in another research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative body movement | During the surgery
  Intraoperative body movement is defined as those likely to interfere with surgical procedures such as bending of hand and/or leg and movement of head.

SECONDARY OUTCOMES:
Neurological function | at discharge and 6 months after operation
  Measured using Markwalder Grading Scale and the Modified Rankin Scale. Markwalder Grading Scale ranges from grade 0 to 4, and the Modified Rankin Scale score ranges from 0 to 6.
Recurrence rate at 6 months after surgery | From operation up to 6 months postoperatively
  Rate of reoperations
Conversion to general anesthesia | During the surgery
  For the nerve block anesthesia combined with sedative anesthesia group, general anesthesia is performed if uncontrolled body movements still exist after opioid and sedative supplement.
Intraoperative awareness | 1 day after surgery
  Measured with the Brice questionnaire. Evaluate Intraoperative awareness through the following 6 questions：1. What is the last thing you remember before going to sleep (please tick one box)?2. What is the first thing you remember after waking up (please tick one box)?3. Do you remember anything between going to sleep and waking up (please tick box)?4. Did you dream during your procedure (please tick box)?5. Were your dreams disturbing to you (please tick box)?6. What was the worst thing about your operation (please tick box)?
Postoperative delirium | 1-5 days after surgery
  POD will be assessed twice a day (before 09:00 and after 16:00) using the Richmond Agitation-Sedation Scale, the Confusion Assessment Method for Intensive Care Unit (CAM-ICU), and the 3- Minute Diagnostic Interview for CAM (3D-CAM).

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Liu, M.D., Principal Investigator — Beijing Tiantan Hospital; Yuming Peng, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong HM, Woo XL, Goh CH, Chee PHC, Adenan AH, Tan PCS, Wong ASH. Chronic Subdural Hematoma Drainage Under Local Anesthesia with Sedation versus General Anesthesia and Its Outcome. World Neurosurg. 2022 Jan;157:e276-e285. doi: 10.1016/j.wneu.2021.10.074. Epub 2021 Oct 11. PMID 34648987
- [Background] Ashry A, Al-Shami H, Gamal M, Salah AM. Local anesthesia versus general anesthesia for evacuation of chronic subdural hematoma in elderly patients above 70 years old. Surg Neurol Int. 2022 Jan 12;13:13. doi: 10.25259/SNI_425_2021. eCollection 2022. PMID 35127213
- [Background] Liu HY, Yang LL, Dai XY, Li ZP. Local anesthesia with sedation and general anesthesia for the treatment of chronic subdural hematoma: a systematic review and meta-analysis. Eur Rev Med Pharmacol Sci. 2022 Mar;26(5):1625-1631. doi: 10.26355/eurrev_202203_28230. PMID 35302209